CLINICAL TRIAL: NCT02029170
Title: Early Weightbearing Versus Non-weightbearing After Operative Treatment of an Ankle Fracture: A Randomized Multicenter Non-inferiority Trial
Brief Title: Early Weightbearing Versus Non-weightbearing After Operative Treatment of an Ankle Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Hyong Nyun Kim, professor, MD, PhD, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUKSHHOS
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Ankle Fracture; Rehabilitation
Keywords: ankle fracture; weightbearing; cast
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early weightbearing (Experimental): After operative reduction and fixation of the fractures, patients allocated to the early weightbearing group start weightbearing after stitch out at 2 weeks and the application of a walking cast.
  Interventions: Procedure: Early weightbearing
- Non-weightbearing (Active Comparator): Patients allocated to non-weightbearing group are kept non-weightbearing till 6 weeks post-operative
  Interventions: Procedure: Non-weightbearing

INTERVENTIONS:
Procedure: Early weightbearing — Patients allocated to early weightbearing group are allowed to weightbear after stitch out and application of a walking cast
  Arms: Early weightbearing
Procedure: Non-weightbearing — Patients allocated to non-weightbearing group are kept non-weightbearing till 6 weeks post-operative
  Arms: Non-weightbearing

SUMMARY:
Unstable ankle fractures are commonly treated operatively. After operative reduction and fixation of the fractures, there are varying rehabilitation regimes that include non-weightbearing for 6 weeks with active range of motion exercise in a removal cast or brace, or early protected weightbearing in a rigid cast. Several papers reported that early weightbearing may decrease ankle stiffness, muscle and bone atrophy, and aids in early return to activities. However, early weightbearing may have the risk of displacement of the fixed fractures. Rehabilitation after operative treatment of an ankle fracture is still not clear. We hypothesized that the ankle function assessed on 12 months after operation of an ankle fracture with early weightbearing is not inferior to non-weightbearing but is superior to non-weightbearing with respect to time to return to normal daily life and time to full weightbearing.

DETAILED DESCRIPTION:
This study is a noninferiority, randomized controlled trial of patients presenting to multiple centers.

The primary outcome measure is the Olerud-Molander scores assess on 12 months after operation of an unstable ankle fracture. The Olerud-Molander scores were compared between the experimental group (early weightbearing) and the control group (non-weightbearing) on 12 month follow-up examination.

The Olerud-Molander score is a most widely used validated scale to assess ankle function after an ankle fracture. It is a self-administered patient questionnaire with a score of zero (totally impaired) to 100 (completely unimpaired) and is based on nine different items: pain, stiffness, swelling, stair climbing, running, jumping, squatting, supports and work/activities of daily living.

The secondary objectives are to determine whether early weightbearing is superior to non-weightbearing with respect to time until return to normal daily life and time to full weightbearing.

Other objectives are to determine safety by assessing number of participants with adverse effect such as hardware failure, reduction loss, non-union, or delayed union in each group.

The sample size was determined using methods appropriate for noninferiority trials, assuming 90% power and a significance level of 0.05. To find out whether the early weightbearing is not inferior to nonweightbearing after operation of an ankle fracture, 192 patients were required to have 90% power that the lower limit of an one-sided 95% confidence interval for the difference between two treatments will be above the noninferiority margin of -8, adding 20% of assumed drop-out.

Determination of the noninferiority margin was based on clinical significance. In a previous study between early weightbearing versus nonweightbearing after an ankle fracture surgery, Simanski et al. reported that both groups showed good results in the Olerud-Molander score (87 vs. 79 points; p=0.25). In both groups, the majority of patients reached their preinjury level of activity. The difference in the Olerud-Molander score between the two groups was 8 points in favor of early weightbearing. Their study came from populations similar to our trial population and from interventions similar to those being studied in the current trial. We decided that the noninferiority margin at 8 points difference will be adequate to prove noninferiority of the experiment group (early weightbearing) over the control group (nonweightbearing).

If a subject had discontinued prior to completion of 12 months, the last observation is carried forward for the intent-to-treat analysis. Subjects who crossed over to the other treatment arm, for an example, patients in non-weightbearing group who weightbear early, are analyzed according to their initial group allocation for the intent-to-treat analysis. Additionally, an as-treated (per-protocal) analysis was also conducted on patients who completed the 12 months follow-up with the protocol assigned.

ELIGIBILITY:
Inclusion Criteria:

* unstable ankle fracture requiring open reduction and internal fixation
* age between 18 and 65 years
* satisfactory reduction and stable fixation after operation.

Exclusion Criteria:

* open fractures
* comminuted fractures
* pathologic fractures
* Pilon fractures
* Trimalleolar fractures
* fracture dislocations
* Fractures requiring syndesmotic screw fixation
* Fractures with cartilage injuries or unstable fixation or any other conditions preventing from early weightbearing.
* Patients with diabetes or neuroarthropathy
* Patients with obesity (BMI >30, weight >100 kg)
* Any other conditions that are expected to prevent the patients from following the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The Olerud-Molander ankle function score | 12 months post-operative
  The Olerud-Molander score is a most widely used validated scale to assess ankle function after an ankle fracture. It is a self-administered patient questionnaire with a score of zero (totally impaired) to 100 (completely unimpaired) and is based on nine different items: pain, stiffness, swelling, stair climbing, running, jumping, squatting, supports and work/activities of daily living.

SECONDARY OUTCOMES:
Time to return to preinjury activity, time to full weightbearing, patients' subjective satisfactions, Visual analogue Scale (VAS) | upto 12 months
  Time to return to preinjury activity and time to full weightbearing is going to be assessed.
  Patient's subjective satisfaction and VAS are going to be assessed on 12 months post-operative visit

OTHER OUTCOMES:
Number of Participants with hardware failure, reduction loss, delayed union or non-union are assessed | Up to 12 month
  A reduction loss or hardware failure was defined as one that occurred without patient instigation of inappropriate activity. The reduction loss or metal failure rate was to be monitored by study personnel not involved in the outcome assessment. >2 mm displacement. Delayed union was defined as a lack of bridging callus on 3 of 5 cortices at 12 weeks. Nonunion was defined as lack of cortical bridging or a clearly visible fracture line, at 14 weeks post injury.

CONTACTS AND LOCATIONS:
Overall Officials: Hyong Nyun Kim, MD, PhD, Study Chair — Kangnam Sacred Heart Hospital, Hallym University College of Medicine; Hyong Nyun Kim, MD, PhD, Study Director — Kangnam Sacred Heart Hospital, Hallym University College of Medicine
Locations (4):
- South Korea (4):
  - Hallym University Sacred Heart Hospital, Hallym University College of Medicine, Anyang-si, Gyeonggi-do
  - Sanbon Hospital, Wonkwang University College of Medicine, Gunpo, Gyeongi
  - CHA Bundang Medical Center, CHA University, Seongnam, Gyeongi
  - Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Seoul

REFERENCES:
- [Background] Ahl T, Dalen N, Holmberg S, Selvik G. Early weight bearing of displaced ankle fractures. Acta Orthop Scand. 1987 Oct;58(5):535-8. doi: 10.3109/17453678709146394. PMID 3425284
- [Background] Aktas S, Kocaoglu B, Gereli A, Nalbantodlu U, Guven O. Incidence of chondral lesions of talar dome in ankle fracture types. Foot Ankle Int. 2008 Mar;29(3):287-92. doi: 10.3113/FAI.2008.0287. PMID 18348824
- [Background] Bostman OM. Body-weight related to loss of reduction of fractures of the distal tibia and ankle. J Bone Joint Surg Br. 1995 Jan;77(1):101-3. PMID 7822361
- [Background] Burwell HN, Charnley AD. The treatment of displaced fractures at the ankle by rigid internal fixation and early joint movement. J Bone Joint Surg Br. 1965 Nov;47(4):634-60. No abstract available. PMID 5846764
- [Background] Dogra AS, Rangan A. Early mobilisation versus immobilisation of surgically treated ankle fractures. Prospective randomised control trial. Injury. 1999 Aug;30(6):417-9. doi: 10.1016/s0020-1383(99)00110-2. PMID 10645355
- [Background] Finsen V, Saetermo R, Kibsgaard L, Farran K, Engebretsen L, Bolz KD, Benum P. Early postoperative weight-bearing and muscle activity in patients who have a fracture of the ankle. J Bone Joint Surg Am. 1989 Jan;71(1):23-7. PMID 2492286
- [Background] Ganesh SP, Pietrobon R, Cecilio WA, Pan D, Lightdale N, Nunley JA. The impact of diabetes on patient outcomes after ankle fracture. J Bone Joint Surg Am. 2005 Aug;87(8):1712-8. doi: 10.2106/JBJS.D.02625. PMID 16085609
- [Background] Lehtonen H, Jarvinen TL, Honkonen S, Nyman M, Vihtonen K, Jarvinen M. Use of a cast compared with a functional ankle brace after operative treatment of an ankle fracture. A prospective, randomized study. J Bone Joint Surg Am. 2003 Feb;85(2):205-11. doi: 10.2106/00004623-200302000-00004. PMID 12571295
- [Background] Mak KH, Chan KM, Leung PC. Ankle fracture treated with the AO principle--an experience with 116 cases. Injury. 1985 Jan;16(4):265-72. doi: 10.1016/s0020-1383(85)80017-6. PMID 3967916
- [Background] Olerud C, Molander H. A scoring scale for symptom evaluation after ankle fracture. Arch Orthop Trauma Surg (1978). 1984;103(3):190-4. doi: 10.1007/BF00435553. PMID 6437370
- [Background] Pagliaro AJ, Michelson JD, Mizel MS. Results of operative fixation of unstable ankle fractures in geriatric patients. Foot Ankle Int. 2001 May;22(5):399-402. doi: 10.1177/107110070102200507. PMID 11428758
- [Background] Simanski CJ, Maegele MG, Lefering R, Lehnen DM, Kawel N, Riess P, Yucel N, Tiling T, Bouillon B. Functional treatment and early weightbearing after an ankle fracture: a prospective study. J Orthop Trauma. 2006 Feb;20(2):108-14. doi: 10.1097/01.bot.0000197701.96954.8c. PMID 16462563
- [Background] Starkweather MP, Collman DR, Schuberth JM. Early protected weightbearing after open reduction internal fixation of ankle fractures. J Foot Ankle Surg. 2012 Sep-Oct;51(5):575-8. doi: 10.1053/j.jfas.2012.05.022. Epub 2012 Jul 20. PMID 22819002
- [Background] Strauss EJ, Frank JB, Walsh M, Koval KJ, Egol KA. Does obesity influence the outcome after the operative treatment of ankle fractures? J Bone Joint Surg Br. 2007 Jun;89(6):794-8. doi: 10.1302/0301-620X.89B6.18356. PMID 17613507
- [Background] Tropp H, Norlin R. Ankle performance after ankle fracture: a randomized study of early mobilization. Foot Ankle Int. 1995 Feb;16(2):79-83. doi: 10.1177/107110079501600205. PMID 7767451
- [Background] Tunturi T, Kemppainen K, Patiala H, Suokas M, Tamminen O, Rokkanen P. Importance of anatomical reduction for subjective recovery after ankle fracture. Acta Orthop Scand. 1983 Aug;54(4):641-7. doi: 10.3109/17453678308992903. PMID 6422695
- [Derived] Park JY, Kim BS, Kim YM, Cho JH, Choi YR, Kim HN. Early Weightbearing Versus Nonweightbearing After Operative Treatment of an Ankle Fracture: A Multicenter, Noninferiority, Randomized Controlled Trial. Am J Sports Med. 2021 Aug;49(10):2689-2696. doi: 10.1177/03635465211026960. Epub 2021 Jul 12. PMID 34251882